CLINICAL TRIAL: NCT05258240
Title: A Randomized Controlled Trial On The Effects Of Virtual Reality-Based Balance Training On Balance In Patients With Diabetic Peripheral Neuropathy
Brief Title: Effects of Virtual Reality-based Balance Training on Balance of Diabetic Peripheral Neuropathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-FSD-00296
Record Dates: First submitted 2022-02-20; First posted 2022-02-28 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Virtual Reality; Balance Training; Balance; Diabetic Peripheral Neuropathy; Randomized Control Trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single-blinded as assessor of the study would be kept blind of the treatment group to which the patient will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Other): Virtual reality workout session will be for about 50 minutes in which warm-up exercise will be for 5 minutes including relaxed breathing, selected exercises for dynamic balance and static balance will take 40 minutes of the session in which games; tilt city, soccer heading, table tilt game, and penguin tilt will be used for dynamic balance training. For static balance training games will be torso leg curl and single leg extension. After that 5 minutes will be given for cools down.
  Interventions: Other: Virtual Reality
- Conventional Physical Therapy (Other): Conventional physical therapy will be provided to this group for 50 minutes, with one minute of rest for every five minutes of exercise. Warm-up for 5 minutes, balancing-drills for 40 minutes, and cools down for five minutes. The session will include; slow and deep breathing exercise for about 3 minutes, patient will be asked to move both ankle joint to its complete range of movement for about five minutes, posture training for balance includes standing from sitting for five times, shifting the weight of the body while standing at one place for five times, move the body to the side and forward to aim the objective set by the therapist for five times, lift or raise the heels for five times of both foot for 20 seconds for each rise, to stand on one foot for 15 seconds, five times, to stand on one foot and bend the knee for about 15 seconds, five times. Wobble board preparation gait training and spot marching will be performed for about 5 to 6 minutes each.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Virtual Reality — Virtual reality workout enhances balance control, self-reported balance and mental stability in healthy and stable adults. Sensory-based exercise and the response to visual acuity can increase the patient's ability to maintain their body in a stable position.
  Arms: Virtual Reality
Other: Conventional Physical Therapy — Postural training, standing, walking, and walking activities are included in the conventional physical therapy in domain of balance exercise training programs. These activities are usually boring and tedious because these exercises are repeated many times.
  Arms: Conventional Physical Therapy

SUMMARY:
The study aimed to clarify the effect of virtual reality-based balance training on balance in patients with diabetic peripheral neuropathy compared to conventional physical therapy.

DETAILED DESCRIPTION:
A randomized control trial will be conducted at the study setting Safi Hospital Faisalabad after the approval of the synopsis. The study will be a single-blinded randomized control study. A convenient sampling technique will be used for the enrollment of the patient. Patient selection will be done based on defined insertion and omission criteria.

Two groups would be made, the intervention group would receive the virtual gaming exercise tutoring and the control group would receive the regular physiotherapy exercises.

The evaluation of the patients will be done at the start of the study, after six weeks, and after twelve weeks. Follow-up will be in the 16th weeks after the cessation of therapy.

The patient's outcome will be measured on Berg Balance Scale and the Single Leg Stance test and the patient's data will be recorded before and after treatment, comparisons between before the treatment and after the treatment data will be made after 12 weeks. Informed consent/approval would be taken from each patient. Analysis and entry of data will be done by Statistical Package of Social Sciences Version 22 Software.

ELIGIBILITY:
Inclusion Criteria:

* Adults age (45-65 years)
* Male and female (both gender)
* Medical diagnoses of type-II diabetes
* DPN confirmed by physician
* Stages ( Ia - sign but no symptoms of neuropathy, Ib - symptomatic mild diabetic poly neuropathy, sensory, motor or autonomic symptoms; patient able to heel walk)
* Patients independent in transfer.
* Unimpaired cognition/intelligence (Mini Mental State Examination Score of >24)

Exclusion Criteria:

* Any neurological diseases e.g. Dementia, Parkinson, Stroke
* Severe visual impairment and Cardiopulmonary disease
* Musculoskeletal disorder, any disease due to individual were unable to walk and lower limb amputation
* Disease which has chances of falling

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | 12th Week
  The Berg Balance Scale is used to objectively determine a patient's ability or inability to safely balance during a series of predetermined tasks. Berg Balance Scale (BBS) is a 14-item objective measure that assesses static balance and fall risk in adults. Berg balance scale scoring ranges from 0 to 56. The lower your score, the more at risk you are for losing your balance. In general, Berg balance scale scores are interpreted as such: 0 to 20: A person with a score in this range will likely need the assistance of a wheelchair to move around safely.
Single leg standing test | 12th Week
  Single leg standing test used to assess static postural and balance control. ... Client must stand unassisted on one leg, timed from the time the other foot leaves the ground till when the foot touches the ground again or the arms leave the hips. Participants unable to perform the one-leg stand for at least 5 seconds are at increased risk for injurious fall.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No